CLINICAL TRIAL: NCT02473900
Title: An Open-label, Randomized, Single-dose Crossover Study to Evaluate the Pharmacokinetics of HIP1403 in Healthy Male Subjects
Brief Title: Evaluating the Bioequivalence of HIP1403, HGP0919
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Hanmi Pharmaceutical Company Limited (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: HM-OSTA-101
Record Dates: First submitted 2015-06-14; First posted 2015-06-17 (Estimated); Last update posted 2016-10-13 (Estimated); Status verified 2016-10

CONDITIONS: Healthy
MeSH Terms: interventions — Oseltamivir

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Sequence 1 (Experimental): HIP1403→HGP0919
  Interventions: Drug: HIP1403; Drug: HGP0919
- Sequence 2 (Experimental): HGP0919→HIP1403
  Interventions: Drug: HIP1403; Drug: HGP0919

INTERVENTIONS:
Drug: HIP1403 — Oseltamivir 75mg
  Other Names: Oseltamivir 75mg
Drug: HGP0919 — Oseltamivir phosphate 75mg
  Other Names: Tamiflu 75mg

SUMMARY:
The purpose of this study is to investigate the bioequivalence after administration of HIP1403 and HGP0919 in healthy male volunteers

DETAILED DESCRIPTION:
A randomized, open-label, single dose, crossover clinical trial to investigate and compare the pharmacokinetics between HIP1403 and HGP0919 in healthy male volunteers.

ELIGIBILITY:
Inclusion Criteria:

1. Healthy male volunteers, age 19 to 45 years.
2. The result of Body Mass Index(BMI) is not less than 18 kg/m2 , no more than 27 kg/m2
3. Subjects who have ability to comprehend the objectives, contents of study and property of study drug before participating in trial and have willingness to sign of informed consent in writing

Exclusion Criteria:

1.Presence of medical history or a concurrent disease that may interfere with treatment and safety assessment or completion of this clinical study, including clinically significant disorders in kidney, liver, cardiovascular system, respiratory system, endocrine system, or neuropsychiatric system.

Ages: 19 Years to 45 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 32 (Actual)
Dates: Start 2015-04; Primary Completion 2015-04 (Actual); Study Completion 2015-04 (Actual)

PRIMARY OUTCOMES:
Oseltamivir Cmax, AUClast , AUCinf | 0h(predose), 0.25, 0.5, 0.75, 1, 1.5, 2, 3, 4, 6, 7, 8, 10, 12, 24, 48hours (Total 16)

SECONDARY OUTCOMES:
Oseltamivir Tmax | 0h(predose), 0.25, 0.5, 0.75, 1, 1.5, 2, 3, 4, 6, 7, 8, 10, 12, 24, 48hours (Total 16)
Oseltamivir t1/2 | 0h(predose), 0.25, 0.5, 0.75, 1, 1.5, 2, 3, 4, 6, 7, 8, 10, 12, 24, 48hours (Total 16)
Oseltamivir CL/F | 0h(predose), 0.25, 0.5, 0.75, 1, 1.5, 2, 3, 4, 6, 7, 8, 10, 12, 24, 48hours (Total 16)
Oseltamivir Vd/F | 0h(predose), 0.25, 0.5, 0.75, 1, 1.5, 2, 3, 4, 6, 7, 8, 10, 12, 24, 48hours (Total 16)

CONTACTS AND LOCATIONS:
Overall Officials: Ji Young Park, MD, PhD, Principal Investigator — Korea University Anam Hospital
Locations (1):
- Korea University Anam Hospital, Seoul, South Korea

IPD SHARING:
Plan to Share IPD: No